CLINICAL TRIAL: NCT05652738
Title: The Impact of Passive Cooling Versus Blanket-Roll III on The Myocardial Function of Asphyxiated Neonates: A Randomized Clinical Trial
Brief Title: Passive Cooling Versus Blanket-Roll III on The Myocardial Function of Asphyxiated Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Primary Investigator and Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0107176
Record Dates: First submitted 2022-11-25; First posted 2022-12-15 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Hypoxic Encephalopathy; Birth Asphyxia; Neonatal Encephalopathy; Hypothermia, Newborn
Keywords: therapeutic hypothermia; asphyxiated neonates; tissue Doppler
MeSH Terms: conditions — Hypoxia, Brain; Asphyxia Neonatorum; Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I: (passive cooling group) (Active Comparator)
  Interventions: Device: Passive cooling application
- Group II: (Blanket roll III cooling group) (Placebo Comparator)
  Interventions: Device: cooling using Blanket roll III

INTERVENTIONS:
Device: Passive cooling application — Passive cooling application for asphyxiated neonates and their effect on myocardial function and hemodynamics
  Arms: Group I: (passive cooling group)
Device: cooling using Blanket roll III — standard care using Blanket roll III in asphyxiated neonates and their effect on myocardial function and hemodynamics
  Arms: Group II: (Blanket roll III cooling group)

SUMMARY:
Studying the effect of passive versus Blanket roll III modality of therapeutic hypothermia (TH)on myocardial function of asphyxiated neonates through using tissue Doppler (TD).

DETAILED DESCRIPTION:
A clinical trial study of 100 Gestational-age-matched asphyxiated cooled neonates will divided into two groups, 50 in each group for comparison the myocardial function using passive cooling and BLANKET ROLL III as modality of TH.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of perinatal/intrapartum hypoxia, as indicated by at least one of:

  * Apgar score of less than or equal to 5 at 10 minutes
  * Needing mechanical ventilation or ongoing resuscitation at 10 minutes
  * PH in cord blood gas is less than 7.00 or a base excess worse than or equal to minus 12 mmol /L on cord/arterial/venous/capillary blood gas obtained within 60 minutes of birth.
* Evidence of moderate or severe encephalopathy.
* Greater than or equal to 35 weeks gestational age.
* Birth weight greater than or equal to 1800 g.
* Able to begin cooling before 6 hours of birth.

Exclusion Criteria:

* Congenital cyanotic heart disease.
* Multiple congenital anomalies.
* Birth asphyxia's babies after start of cooling with cardiovascular instability.

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Myocardial function through using tissue Doppler (TD). | first 4 days of life
  neonatal echocardiography using a (Vivid IQ) with a (3-8 MHz) with software for Tissue Doppler imaging (TDI) , myocardial performance index and measuring velocities of different waveforms, cm/sec.
Left ventricular function through using conventional echocardiography. | first 4 days of life
  Ejection fraction in percent .

SECONDARY OUTCOMES:
Right ventricular function using conventional echocardiography | first 4 days of life
  TAPSE (tricuspid annular plane systolic excursion) in mm .

CONTACTS AND LOCATIONS:
Overall Officials: Reham M Wagdy, PhD, Principal Investigator — Faculty of medicine, Alexandria University, Egypt; Hossam M Kamel, MBChB, Principal Investigator — Faculty of medicine, Alexandria University, Egypt; Rasha M Adel Nasra, Principal Investigator — Alexandria University
Locations (1):
- Marwa Mohamed Farag, Alexandria, Egypt